CLINICAL TRIAL: NCT03098095
Title: The Use of a Mobile Application to Support Physical Activity and Lifestyle Changes in Persons Living With HIV: the SMARTAPP Study.
Brief Title: A Smartphone Application to Support Physical Activity in HIV Infected People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Collaborators: University of Milan (Other); Catholic University of the Sacred Heart (Other); IRCCS Lazzaro Spallanzani (Unknown); University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Paola Cinque, Medical Doctor, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSR - Prot. SMARTAPP
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Physical Activity; HIV Infections
MeSH Terms: conditions — Motor Activity; HIV Infections | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Open-Label, Randomized, Multicenter, Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Device smartphone. Participants will be trained with a supervised physical activity for 3 days a week for 16 weeks with the use of a smartphone application
  Interventions: Behavioral: Physical Activity
- Control Group (Experimental): Participants will train alone with an exercise program for 16 weeks without the use of a smartphone application
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Moderate physical activity

SUMMARY:
Physical activity delays all-cause mortality in the general population and reduces the risk of cardiovascular disease (CVD), stroke, type-2 diabetes and some types of cancer (Garber et al., 2011). These diseases are associated with chronic inflammation, which is characterized by activation of inflammatory signalling pathways with abnormal production of cytokines and other mediators (Hotamisligil, 2006). Observational studies of large population cohorts have consistently shown an association between physical inactivity and low-grade systemic inflammation and interventional studies a reduction of inflammatory markers following exercise (Beavers et al., 2010).

Chronic inflammation is also a predominant feature of treated human immunodeficiency virus (HIV) infection (Lederman et al., 2013; Deeks et al., 2013). Compared to age-matched HIV-negative subjects, persons with chronic HIV infection are at higher risk to develop non-acquired immune deficiency syndrome (AIDS) related chronic diseases (Guaraldi et al., 2011), and several studies have shown an association between chronic inflammation and higher cardiovascular risk and overall mortality (Kuller et al., 2008, Duprez et al., 2012).

Recently, the investigators performed a pilot study of moderate physical activity that enrolled sedentary HIV infected subjects treated with combination antiretroviral treatment (cART), consisting of brisk walking, with or without strength exercise. Overall, after 12 weeks of training cholesterol profile and soluble and cell inflammatory markers improved significantly. However, because of the considerable individual variability in exercise responses, a program of physical activity needs be adjusted on an individual basis to be most effective. During recent years, the use of mobile technologies has been implemented for health monitoring interventions, including exercise. We hypothesized that the use of a mobile application will favour engagement to exercise by providing motivational inputs, and therefore adherence, and, as a consequence, an improvement of physical fitness.

The investigators hypothesized that the use of a mobile application will favour engagement to exercise by providing motivational inputs, and therefore adherence, and, as a consequence, an improvement of physical fitness. Therefore, the aim of this project is to improve health and quality of life of patients living with HIV through self-empowerment by use of an innovative mobile application, in order to assist and monitor individualized program of physical activity and diet recommendation.

OBJECTIVES

Primary To compare the improvement of physical fitness between the EG and CG groups after 16 weeks of training.

Secondary

To compare the improvement of the following characteristics between the EG and CG groups after 16 weeks of training:

1. anthropometry,
2. Blood lipids,
3. Inflammatory markers,
4. Quality of Life,

4. Mood State.

ENDPOINTS Primary The primary objective will be assessed by the proportion of subjects with an improvement from baseline of 15% of maximal oxygen consumption (O2max) through 16 weeks of training.

Secondary

The secondary endpoints will be assessed by the 16-week changes in the following measures:

1. BMI and %Fat Mass,
2. Blood Total-, LDL-, HDL-Cholesterol,
3. Blood IL-6, hs-PCR, d-Dimer, IL-18; myostatin; T-cell activation markers,
4. F12 questionnaire,
5. Profile of Mood State questionnaire.

DETAILED DESCRIPTION:
STUDY DESIGN Multicentre, randomized, open-label, pilot study enrolling HIV-infected subjects, of age ≥18 years, with or without cART, either sedentary or already practicing mild/moderate physical activity.+

Subjects satisfying the inclusion and exclusion criteria will be randomized 1:1 to one of the following arms:

i) experimental group (EG), where participants will be trained with an exercise program for 16 weeks with the use of a smartphone application; ii) control group (CG), where participants will be trained with an exercise program for 16 weeks without smartphone application.

You will be screened for eligibility by an infectious diseases specialist and a sport medicine specialist through collection of clinical and treatment history, physical examination, routine blood screen, ECG at rest and during submaximal cycle ergometer test. Eligible patients will sign a written informed consent and will be followed-up at screening, baseline (start of the training program) and after 16 weeks of training, except for profile of mood states that will be assessed weekly

Each study visit will include: the evaluation of CDC stage, anthropometric assessment (height, weight), systolic and diastolic blood pressure, smoking status, assessment of the antiretroviral and concomitant therapies and routine laboratory tests. Additional 30 mL of peripheral blood will be withdrawn at baseline and at the end of the study (week 16) and stored in a biobank for further investigations for patients recruited from San Raffaele Hospital. The demographic, clinical, physical fitness, quality of life information will be accurately recorded at the study visits in an electronic Case Report Form (eCRF).

Randomization Randomization list will be computer-generated (block sizes of ten) and will be incorporated within the electronic clinical report form (eCRF) of the study. Study participants, study nurses and study physicians will be aware of the allocation group but allocation will be concealed from laboratory staff.

Discontinuation from the study You may withdraw consent at any time for any reason or be dropped from the study at discretion of the investigator if he/she violates the study plan or for administrative or other reasons.

You will be discontinued from the study if you will:

* withdraw consent or
* miss the exercise sessions for ≥ 2 consecutive weeks (corresponding to 6 sessions).

Any female patient who becomes pregnant during the course of the study will be also immediately withdrawn from the study.

Exercise program The exercise prescription will be scheduled according to the American College of Sport Medicine guidelines (Garber et al., 2011). You will perform 3 outdoor training sessions a week for 16 weeks, consisting of brisk walking or running for one hour. In both groups, participants will be assigned the same volume and intensity of exercise. After baseline O2max examination, participants will receive and individual training program written by exercise scientists (MB, GP, ALT), which will be designed according to the performance at O2max examination. The exercise program will be divided into two periods. In the first period (weeks 1-4) subjects will train at 60-70% of maximal heart rate to improve the aerobic metabolism capacity. Moreover, participants will be familiarized to both physical activity (both EG and CG) and the use of mobile application (the EG only) through direct coach supervision. In the second period (weeks 5-16), participants will train without direct coach supervision, but following the individualized program on a designed timeline. The EG participants will receive automatic real-time feedback though the application and both EG and CG participants weekly feed-back from trainers. During this period exercise intensity, will be increased to 70-80% of maximal heart rate.

Training adherence Adherence to the program will be defined as the proportion of sessions attended during the 16-week training period and it will be calculated only among the participants who will complete the study.

Anthropometric Assessment The anthropometric assessment will be performed before and at the end of the program by the same operator following the standardized techniques described by Lohman (1981). Anthropometric variables will include body mass, stature, and skinfold thickness on the dominant side. Stature and body mass will be measured with a portable stadiometer and scaled to the nearest 0.5 cm and 0.1 kg, respectively. Skinfolds will be taken three times in each anatomic site using a calliper (Holtain Ltd, Crymych Uk) to the nearest 0.2 mm. The average value obtained among the three measures will be computed. Body density (d) will be calculated using the Jackson & Pollock equation (1985) from three skinfolds (Female: triceps, suprailiac and thigh; Male: pectoral, abdominal and thigh). The percentage of fat mass will be finally derived as: fat mass (%) = 495/ d - 450 (Siri et al., 1961).

Physical Fitness Evaluation You will be instructed to arrive at the laboratory in a rested and fully hydrated state and to avoid strenuous exercise in the 24 h preceding the testing session. In addition, they will avoid alcohol intake in the 48 h before the exercise test. All tests will be carried out in a well-ventilated laboratory at a temperature of 20-22°C on an electromagnetically-braked cycle ergometer (Monarc, Ergometric 893, Finland). The protocol will begin with subjects cycling at 50 W for 6 minutes; then the load will increase by 15 W each minute until volitional exhaustion. The peak values of the main cardiovascular, respiratory, and metabolic parameters will be taken as the highest 30-s mean value attained before the subject's volitional exhaustion. Oxygen consumption (), carbon dioxide production (), respiratory exchange ratio (RER) and pulmonary ventilation () will be measured on a breath-by-breath basis by telemetric metabolimeter (Quarkb2, Cosmed, Rome, Italy). O2max will be assessed according to the criterion described by Taylor et al. Heart rate (HR) will be recorded during the whole test by a HR monitor (Polar S810, © Polar Electro 2011, Kempele, Finland). The VT will be assessed according to the gas exchange method (V-Slope).24 Briefly, the break point in the vs relationship will be detected and considered as the VT. Then the VT will be expressed in percentage of the max.

Rating of Perceived Exertion The Borg 6-20 scale is selected to rate the perceived intensity of exertion (Borg, 1982). A verbal-anchored scale will be shown to participants before, immediately and after 30-min completing the training session. Each subject will be familiarized on the use of Borg 6-20 scale, including anchoring procedures.

Total Quality Recovery scale (TQR) Psychophysiological recovery process status will be checked using the Total Quality Recovery scale (TQR) (Kenttä et al., 1998). Participants will provide a rating of perceived quality of recovery using a scaling from 6 (worst) to 20 (best). A verbal-anchored scale will be shown to the subjects, the morning after the training session. Each subject will be familiarized on the use TQR scale, including anchoring procedures.

Profile of Mood State (POMS) The POMS questionnaire contains 32 items reflecting an individual's mood on five primary dimensions (i.e. depression, fatigue, vigour, tension and anger). Subjects will complete POMS individually once a week. The POMS data will be analysed for each specific dimension and "energy index" was calculated as "vigour-fatigue" and used to monitor changes in energy balance.

Quality of life The SF-12 questionnaire is derived from Short-Form Health Survey (36-item). It is a patient-reported survey of patient health (Brazier et al., 1992). This questionnaire was used to evaluate the participant's perception of QOL in the domains of physical functioning, role limitations due to physical health, emotional well-being, social functioning and general health with higher scores indicating greater QOL.

Nutrition The use of a daily food diary will be adopted to assess the nutritional habits of participants; the diary will be fulfilled at least 3 days a week (during 2 working days and 1 day during week-end) and the patient will be requested to indicate the name, the amount and the cooking method of consumed foods and seasonings; beverages will also be included in the report. Diet quality and diet variety indexes will be evaluated starting from the food diary provided by the patients.

Concomitant medications The use of concomitant medications/therapies (already ongoing or that might need to be prescribed during the study) are allowed and recorded. No specific restrictions are foreseen during the course of the study with regard to concomitant therapy or vaccination.

Laboratory analysis Blood examination will include complete blood count; standard biochemical exams with fasting total, high-density lipoprotein (HDL) and low-density lipoprotein (LDL) cholesterol, triglycerides, glucose, insulin, glycated haemoglobin (HbA1c); cluster of differentiation 4 (CD4+) and cluster of differentiation 8 (CD8+) T-cell counts, HIV-1-RNA plasma level (Abbott RealTime HIV-1 assay). The Homeostatic Model Assessment (HOMA)-I and the Veterans Aging Cohort Study Risk (VACS) indexes will also be calculated [15].

Inflammatory markers Soluble biomarkers will be measured in cryopreserved plasma samples, drawn at BL and at the end of the program, by commercially available enzyme-linked immunosorbent assays according to manufacturers' recommendation. These will include high-sensitivity C-reactive protein (hsCRP, Catalog Number DCRP00), interleukin-6 (IL-6, Catalog Number D6050), D-dimer (Asserachrom, Diagnostica Stago, Asnieres-Sur-Seine, France), interleukin-18 (IL-18) (Medical and Biological Laboratories, Nagoya, Japan), myostatin (Cusabio, China).

Flow cytometry for cell-activation markers will be measured on cryopreserved peripheral blood mononuclear cells isolated by Ficoll-Paque gradient from EDTA-anticoagulated whole blood. After thawing and PBS-washing, 3 x 105 cells will be stained using phycoerythrin (PE)-conjugated anti-HLA-DR, PE-cyanin red 5.1-conjugated anti-CD38, Alexa Fluor 647-conjugated anti-CD3, fluorescein isothiocyanate-conjugated anti-CD4 or anti-CD8 (BD-Biosciences, San Diego, CA). CD38+ and HLA-DR+ cells will be gated from the CD3+/CD4+ or CD3+/CD8+ cells on a 2-dimensional dot plot. Analyses will be performed by FACSCalibur with CellQuest software (BD-Biosciences) and results reported as percentages of CD3+/CD4+ and CD3+/CD8+ T-cells expressing both HLA-DR and CD38.

For both soluble and inflammatory markers, samples will be analysed in batch at the end of the study and blindly with respect to group assignment.

Sample size We estimated that a sample size of 48 patients per group, or a total of 96 subjects would be required in order to detect a 30% increase in the proportion of subjects with an improvement of VO2max through 16 weeks of training, from 40% (hypothesized for the control arm, i.e. no use of the smartphone application) to 70% (hypothesized for the experimental arm, i.e. use of the smartphone application arm), with 80% power at an α of 0.05.

As the improvement of VO2max is directly correlated to the adherence to training sessions, we expect that the proportion in the experimental arm (using the smartphone application as supervision) might be similar to that observed in a previous paper (Bonato et al., 2016), reporting that the adherence to exercise program with the supervision of professional coaches was found to be 67%. On the contrary, in absence of training supervision (control group) we expect a lower adherence, i.e. 40%. As the accrual of such a number of subjects is not feasible, we plan to enrol 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* with or without cART;
* either sedentary or already practicing mild/moderate physical activity;

Exclusion Criteria:

* any disease requiring hospitalization in the 6 weeks before enrolment;
* medical conditions contraindicating exercise as established by a sport medicine specialist;
* current substance or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Physical Fitness | After 16 weeks of training
  Improvement of 15% of maximal oxygen consumption

SECONDARY OUTCOMES:
Anthropometry | After 16 weeks of training
  BMI in kg/m^2, weight in kilograms, height in meters
Anthropometry | After 16 weeks of training
  Fat Mass in percentage
Blood Lipids | After 16 weeks of training
  Total cholesterol mg/dL^1
Blood Lipids | After 16 weeks of training
  LDL cholesterol, mg/dL^1
Blood Lipids | After 16 weeks of training
  HDL cholesterol mg/dL^1
Inflammatory Markers | After 16 weeks of training
  Changes of IL-6, IL-18, hs-CRP, d-Dimer, myostatin, T-cell activation markers
Mood States | After 16 weeks of training
  Changes of mood states assessed by Profile of Mood States Questionnairre

OTHER OUTCOMES:
Life quality | After 16 weeks of training
  Changes of quality of life by F12 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonato M, Galli L, Passeri L, Longo V, Pavei G, Bossolasco S, Bertocchi C, Cernuschi M, Balconi G, Merati G, Lazzarin A, La Torre A, Cinque P. A pilot study of brisk walking in sedentary combination antiretroviral treatement (cART)- treated patients: benefit on soluble and cell inflammatory markers. BMC Infect Dis. 2017 Jan 11;17(1):61. doi: 10.1186/s12879-016-2095-9. PMID 28077069